CLINICAL TRIAL: NCT03799848
Title: Phase 1, Open-Label, Parallel-Group, Pharmacokinetic Single Dose Study of Oral Vadadustat in Subjects With Normal and Impaired Hepatic Function
Brief Title: A Single Dose Study of Oral Vadadustat in Subjects With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AKB-6548-CI-0024
Record Dates: First submitted 2018-12-27; First posted 2019-01-10 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Healthy subjects; Child-pugh; Vadadustat
MeSH Terms: interventions — vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vadadustat (Experimental): Group 1: Subjects with moderately impaired hepatic function (Child-Pugh Class B) Group 2: Normal healthy volunteers Group 3: Subjects with mildly impaired hepatic function (Child-Pugh Class A)
  Interventions: Drug: Vadadustat

INTERVENTIONS:
Drug: Vadadustat — Oral tablet
  Other Names: AKB-6548

SUMMARY:
This is a Phase I open-label study to evaluate the pharmacokinetic (PK) profile of a single oral dose of vadadustat in subjects with hepatic impairment(HI) compared to healthy matched control subjects with normal hepatic function.

DETAILED DESCRIPTION:
This is an open label, parallel-group, single dose, Phase 1 study to evaluate the PK profile, safety, and tolerability of a single oral 450 mg dose of vadadustat in subjects with hepatic impairment relative to control subjects with normal hepatic function. The study will enroll up to 24 subjects in 3 groups of 8 subjects at 2 study sites. Blood samples for vadadustat PK and its metabolites will be collected pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 60, and 72 hours post-dose.

ELIGIBILITY:
Inclusion Criteria (All groups):

* Male or female subjects between ≥18 years and ≤70 years of age
* Have a body weight ≥45 kg and body mass index (BMI) ≥18.5 kg/m2 to 40.0 kg/m2

Additional Group-Specific Inclusion Criteria:

* Group 1 (Moderate Hepatic Impairment Subjects):

  * Presence of Moderate hepatic impairment (Child-Pugh Class B)
* Group 2 (Normal Hepatic Function Subjects):

  * Normal hepatic function
* Group 3 (Mild Hepatic Impairment Subjects):

  * Presence of mild hepatic impairment ( Child-Pugh Class A)

Exclusion Criteria (all groups):

* Renal impairment ≥ Stage 3 (estimated glomerular filtration rate [eGFR] <60 mL/min/1.73m2 using the Modification of Diet in Renal Disease (MDRD) study equation)
* Any history of active malignancy within 2 years prior to or during screening, except for treated basal cell carcinoma of skin, curatively resected squamous cell carcinoma of skin, or cervical carcinoma in situ; any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive test for human immunodeficiency virus (HIV) antibody at Screening.
* Hepatic or other organ or cell transplant
* Subjects with alcoholic cirrhosis must be sober for a minimum of 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from dosing to last measurable concentration (AUClast) | Day 1, Day 4
Area under the concentration-time curve from dosing to infinity (AUCinf) | Day 1, Day 4
Observed maximum concentration (Cmax). | Day 1, Day 4

SECONDARY OUTCOMES:
Time to reach Cmax of vadadustat | Day 1, Day 4
Apparent total body clearance (CL/F) of vadadustat | Day 1, Day 4
Apparent volume of distribution (Vd/F) of vadadustat | Day 1, Day 4
Terminal half-life (t1/2) of vadadustat | Day 1, Day 4
Time to reach Tmax of vadadustat | Day 1, Day 4
Assessment of Treatment-Emergent Adverse Events (TEAEs) as reported by study subjects | Up to 9 Weeks
Cmax related to free drug (Cmax, free) of Vadadustat Unbound | Day 1, Day 4
AUClast related to free drug (AUClast, free) of Vadadustat Unbound | Day 1, Day 4
AUCinf related to free drug (AUCinf, free) of Vadadustat Unbound | Day 1, Day 4
CL/F related to free drug (CL/Ffree) of Vadadustat Unbound | Day 1, Day 4
Terminal half-life (t1/2) of Vadadustat Unbound | Day 1, Day 4
The area under the concentration-time curve from dosing to last measurable concentration (AUClast) of Vadadustat metabolites | Day 1, Day 4
The area under the concentration-time curve from dosing to infinity (AUCinf) of Vadadustat metabolite | Day 1, Day 4
Time to reach Cmax of vadadustat metabolites | Day 1, Day 4
Terminal half-life (t1/2) of Vadadustat metabolites | Day 1, Day 4
Renal clearance (CLr) of Vadadustat/metabolite(s) Urine | Day 1, Day 4
Cumulative amount of drug excreted (Ae) of Vadadustat/metabolite(s) Urine | Day 1, Day 4
Cumulative fraction of drug excreted (Fe) of Vadadustat/metabolite(s) Urine | Day 1, Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Akebia Therapeutics
Locations (2):
- United States (2):
  - Prism Clinical Research, Saint Paul, Minnesota
  - American Research Corporation at the University of Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided